CLINICAL TRIAL: NCT06247462
Title: Ibuprofen and Biomarkers of Acute Kidney Injury After Running in the Heat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IBU2023
Record Dates: First submitted 2023-12-19; First posted 2024-02-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ibuprofen (Experimental): 600 mg of Ibuprofen was ingested 12- and 1-hour prior to exercise.
  Interventions: Drug: Ibuprofen 600 mg
- Placebo (Corn Starch) (Placebo Comparator): 600 mg of corn starch was ingested 12- and 1-hour prior to exercise.
  Interventions: Drug: Placebo Corn Starch

INTERVENTIONS:
Drug: Ibuprofen 600 mg — 600 mg of ibuprofen was ingested 12- and 1-hours prior to exercise.
  Arms: Ibuprofen
Drug: Placebo Corn Starch — 600 mg of corn starch (placebo) was ingested 12- and 1-hours prior to exercise.
  Arms: Placebo (Corn Starch)

SUMMARY:
The goal of this study is to determine if ibuprofen prior to exercise in the heat worsens biomarkers of acute kidney injury. Participants were given 600mg of ibuprofen or placebo (corn starch) 12- and 1-hour prior to running for 1-hour in a hot environment (35°C) at moderate intensity. Urine, plasma, and serum samples were collected pre-, post-, and 1hour post-exercise to assess biomarkers of acute kidney injury. This was a double blind, randomized crossover design, so that participants completed the alternate trial (ibuprofen or placebo) at least seven days later.

ELIGIBILITY:
Inclusion Criteria:

* Physically active (engage in at least 150 minutes of moderate to vigorous intensity exercise per week)
* between the ages of 18 and 45
* Able to run continuously for at least 60 minutes
* Able to speak and read English.

Exclusion Criteria:

* Non-English speakers, prisoners, pregnant women, or persons requiring a LAR
* Previous history of heat stroke or heat illness
* Currently experiencing a sunburn or other burn injury
* Have repeated exposure to heat, such as hot baths, sauna, or travel to a hot environment
* Has resided in a hot climate within 2 months prior to the trial
* Answered "yes" to at least one question on the physical activity readiness questionnaire
* Shows signs or symptoms of or are known to have cardiovascular, renal, metabolic, or pulmonary disease as determined by a health questionnaire
* Are a current smoker
* History of regular gastrointestinal distress
* Known history of stomach ulcers or taking blood thinning medication
* Known allergy to ibuprofen
* Have a resting blood pressure greater than 140 systolic or 90 diastolic
* Do not engage in at least 150 minutes of moderate to vigorous intensity exercise per week.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Biomarker of Acute Kidney Injury Risk from Ibuprofen Ingestion Prior to Exercise in the Heat (IGFBP7xTIMP2) | Change in urinary IGFBP7xTIMP2 pre-exercise and 1 hour post-exercise.
  The product of urinary IGFBP7 and urinary TIMP2 (IGFBP7xTIMP2) will be measured at all time points.
Biomarker of Acute Kidney Injury Risk from Ibuprofen Ingestion Prior to Exercise in the Heat (Urinary NGAL) | Change in urinary NGAL pre-exercise and peak post-exercise.
  Urinary NGAL will be measured at all time points.
Biomarker of glomerular filtration rate from Ibuprofen Ingestion Prior to Exercise in the Heat (Serum cystatin C) | Change in serum cystatin C pre-exercise and 1 hour post-exercise.
  Serum cystatin C will be measured at all time points.

SECONDARY OUTCOMES:
Circulating Marker of Intestinal Injury from Ibuprofen Ingestion Prior to Exercise in the Heat | Change in plasma I-FABP from pre- to immediately 1 hour post-exercise.
  Plasma I-FABP is a circulating marker of intestinal damage.
Circulating Marker of Intestinal Permeability from Ibuprofen Ingestion Prior to Exercise in the Heat | Change in plasma LBP from pre- to immediately 1 hour post-exercise.
  Plasma LBP is a circulating marker of intestinal permeability.
Circulating Marker of Endotoxemia from Ibuprofen Ingestion Prior to Exercise in the Heat | Change in plasma sCD14 from pre- to immediately 1 hour post-exercise.
  Plasma sCD14 is a circulating marker of endotoxemia.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Physiology Lab, Albuquerque, New Mexico, United States